CLINICAL TRIAL: NCT05531890
Title: Crossover Study to Evaluate the Comparative Bioavailability, Pharmacokinetics, and Safety of GTX-102 Administered as an Oral Spray Compared to Intramuscular Injection and an Oral Solution of Betamethasone in Healthy Subjects
Brief Title: Comparative Bioavailability of Betamethasone Oral Solution Metered Spray (GTX-102) in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grace Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GTX-102-001
Record Dates: First submitted 2022-08-31; First posted 2022-09-08 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-06

CONDITIONS: Ataxia Telangiectasia
MeSH Terms: conditions — Ataxia Telangiectasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1 GTX-102 medium dose fast or slow in Period 1 and Period 2 (Experimental): GTX-102 Betamethasone oral spray medium dose (0.05 mg/kg) administered fast or slow over two periods
  Interventions: Drug: GTX-102 medium dose fast Period 1 and Period 2; Drug: GTX-102 medium dose slow Period 1 and Period 2
- Group 2a GTX-102 high dose fast in Period 1 and Period 2 (Experimental): GTX-102 Betamethasone oral spray high dose (0.1 mg/kg) administered fast over two periods
  Note: Note under US IND
  Interventions: Drug: GTX-102 high dose fast Period 1 and Period 2
- Group 2b Oral comparator in Period 1 and Period 2 (Active Comparator): 0.1 mg/kg betamethasone solution oral drops solution over two periods
  Note: Not under US IND
  Interventions: Drug: Betamethasone Oral Solution Period 1 and Period 2
- Group 3 GTX-102 high dose fast or low dose fast in Period 1 and Period 2 (Experimental): GTX-102 Betamethasone oral spray high dose (0.1 mg/kg) or GTX-102 Betamethasone oral spray low dose (0.025 mg/kg) administered fast over two periods
  Interventions: Drug: GTX-102 high dose fast Period 1 and Period 2; Drug: GTX-102 low dose fast Period 1 and Period 2
- Group 4a GTX-102 high dose fast in Period 1 and Period 2 (Experimental): GTX-102 Betamethasone oral spray high dose (0.1 mg/kg) administered fast over two periods
  Interventions: Drug: GTX-102 high dose fast Period 1 and Period 2
- Group 4b betamethasone intramuscular in Period 1 and Period 2 (Active Comparator): 0.1 mg/kg betamethasone solution as intramuscular injection administered over two periods
  Interventions: Drug: Betamethasone solution as intramuscular injection Period 1 and Period 2

INTERVENTIONS:
Drug: GTX-102 medium dose fast Period 1 and Period 2 — GTX-102 Betamethasone oral spray medium dose (0.05 mg/kg) administered in Period 1 and Period 2 fast
  Arms: Group 1 GTX-102 medium dose fast or slow in Period 1 and Period 2
Drug: GTX-102 medium dose slow Period 1 and Period 2 — GTX-102 Betamethasone oral spray medium dose (0.05 mg/kg) administered in Period 1 and Period 2 slow
  Arms: Group 1 GTX-102 medium dose fast or slow in Period 1 and Period 2
Drug: GTX-102 high dose fast Period 1 and Period 2 — GTX-102 Betamethasone oral spray high dose (0.1 mg/kg) administered in Period 1 and Period 2 fast
  Arms: Group 2a GTX-102 high dose fast in Period 1 and Period 2; Group 3 GTX-102 high dose fast or low dose fast in Period 1 and Period 2; Group 4a GTX-102 high dose fast in Period 1 and Period 2
Drug: GTX-102 low dose fast Period 1 and Period 2 — GTX-102 Betamethasone oral spray high dose (0.025 mg/kg) administered in Period 1 and Period 2 fast
  Arms: Group 3 GTX-102 high dose fast or low dose fast in Period 1 and Period 2
Drug: Betamethasone solution as intramuscular injection Period 1 and Period 2 — reference product 0.1 mg/kg betamethasone solution as an intramuscular injection
  Arms: Group 4b betamethasone intramuscular in Period 1 and Period 2
Drug: Betamethasone Oral Solution Period 1 and Period 2 — Comparator product 0.1 mg/kg betamethasone oral drops solution
  Arms: Group 2b Oral comparator in Period 1 and Period 2

SUMMARY:
A Randomized, Open-label, Crossover Study to Evaluate the Comparative Bioavailability, Pharmacokinetics, and Safety of GTX-102 Administered as an Oral Spray Compared to Intramuscular Injection - betamethasone and an Oral Solution of Betamethasone in Healthy Subjects.

Four groups of subjects will receive 2 treatments each and randomized in 2-way crossover.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects between the ages of 18 and 55 years, inclusive.
2. Willing and able to provide written informed consent prior to participating in the study.
3. Able to communicate clearly with the Investigator and staff; able to read, complete questionnaires, and understand study procedures.
4. Able to complete all screening period evaluations, and stay in the clinic testing facility for up to 2 consecutive days on 2 separate occasions.
5. Body mass index (BMI) between 18 and 32 kg/m2, inclusive, and body weight between 40 and 120 kg, inclusive.

Exclusion Criteria:

1. Has a history of or current clinically significant medical illness including (but not limited to) pulmonary, cardiovascular, coagulation disorders, lipid abnormalities, gastrointestinal, immunologic, endocrine (stable thyroid hormone replacement therapy is not excluded), neurologic, psychiatric, or thromboembolic disease, metabolic disturbances, or any other current physical condition that the Investigator considers should exclude the participant, or that could interfere with the interpretation of the study results.
2. Has current or recent (within 6 months) history of gastrointestinal disease, or any surgical or medical condition such as Crohn's disease or liver disease, that could potentially alter the absorption, metabolism, or excretion of the study drug.
3. Has any clinically significant medical condition, physical examination finding, vital signs, ECG abnormality (at screening), or clinically significant abnormal value for hematology, serology, clinical chemistry, or urinalysis at screening or at admission to the study center, as deemed appropriate by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2023-05-03 (Estimated)

PRIMARY OUTCOMES:
AUC from 0 to 72 hours post-dose | Up to 72 hours post-dose
  Area under the curve
AUC | Up to infinity
  Area under the curve
Cmax from 0 to 72 hours post-dose | Up to 72 hours post-dose
  Maximum concentration

SECONDARY OUTCOMES:
Adverse Events from Day 1 to Day 45 | Day 1 to Day 45
  Adverse events
Relative bioavailability of GTX-102 oral spray versus betamethasone oral solution and betamethasone intramuscular injection | Up to 72 hours post-dose
  Area under the curve (AUC0-t)
Relative bioavailability of GTX-102 oral spray versus betamethasone oral solution and betamethasone intramuscular injection | Up to infinity
  Area under the curve (AUC0-inf)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Faulknor, MD, Principal Investigator — Clinical Research Unit
Locations (1):
- Clinical Research Unit, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No